CLINICAL TRIAL: NCT05661149
Title: Closed-Loop Insulin Delivery in Pregnant Women with Type 1 Diabetes
Brief Title: Closed-Loop Insulin Delivery During Pregnancy (IADIABENCEINTE)
Acronym: IADIABENCEIN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/0036
Record Dates: First submitted 2022-11-21; First posted 2022-12-22 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes
Keywords: artificial pancreas; closed loop insulin delivery; glucose control; pregnancy; type 1 diabetes; observational study
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Hybrid closed loop insulin delivery systems — Tandem Control-IQ ; DBLG1 system ; MiniMed 780G system

SUMMARY:
The imbalance of diabetes is associated with an increased risk of maternal and fetal complications. In women, it can cause abortion, hypertension, preeclampsia, and obstructed labor; in the fetus, it increases the risk of many malformations, including neurological and cardiac, fetal death in utero, intrauterine growth retardation, macrosomia, prematurity and metabolic complications.

Despite the various therapeutic tools available and used during pregnancy, maintaining blood sugar levels within this narrow range remains a challenge.

Automated Insulin Therapy (IA) Could Further Improve Outcomes With Continuous Glucose Monitoring and Increase Percentage of Time Spent on Target Between 63 and 140 mg/dL The objective of this observational study is to describe the clinical characteristics, metabolic data on MCG and maternal and/or fetal complications in women with T1D treated during pregnancy with an AI system available in France.

DETAILED DESCRIPTION:
Diabetes imbalance is associated with an increased risk of maternal and fetal complications, and achieving target blood glucose levels before and during pregnancy in women with type 1 diabetes (T1DM) significantly reduces these complications. In women, it can cause abortion, hypertension, pre-eclampsia, and dystocic deliveries; in the fetus, it increases the risk of numerous malformations, including neurological and cardiac, fetal death in utero, intrauterine growth retardation, macrosomia, prematurity, and metabolic complications at birth such as neonatal hypoglycemia and hypocalcemia.

The recommended glycemic targets during pregnancy are strict: HbA1c < 6.5% and time in target (between 63 and 140 mg/dL) > 70% (6).

Despite the various therapeutic tools available and used during pregnancy, maintaining blood glucose within this narrow range remains a challenge.

Automated insulin therapy (AI) could improve further on the results obtained with continuous glucose monitoring and increase the percentage of time spent in target between 63 and 140 mg/dL The objective of this present observational study is to describe the clinical characteristics, metabolic data on MCG and maternal and/or fetal complications in women with T1DM treated during pregnancy with an AI system available in France, whether this system is used before the beginning of the pregnancy or during it.

ELIGIBILITY:
Inclusion Criteria:

* aged at least 18 years
* had been diagnosed with type 1 diabetes before pregnancy
* using an hybrid closed-loop insulin delivery system before or at any time of pregnancy

Exclusion Criteria:

* Patient opposed to the research

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients followed in the diabetology department of the Centre Hospitalier Sud-Francilien
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Percentage time spent in the euglycaemic range specific for pregnancy (63-140 mg/dL) | 12 weeks before the start of pregnancy (week 0)
  Data drawn from continuous glucose monitoring systems
Percentage time spent in the euglycaemic range specific for pregnancy (63-140 mg/dL) | week 0
  Data drawn from continuous glucose monitoring systems
Percentage time spent in the euglycaemic range specific for pregnancy (63-140 mg/dL) | Week 14
  Data drawn from continuous glucose monitoring systems
Percentage time spent in the euglycaemic range specific for pregnancy (63-140 mg/dL) | Week 26
  Data drawn from continuous glucose monitoring systems
Percentage time spent in the euglycaemic range specific for pregnancy (63-140 mg/dL) | Wekk 38
  Data drawn from continuous glucose monitoring systems

CONTACTS AND LOCATIONS:
Overall Officials: Alfred PENFRONIS, PHD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France, France

IPD SHARING:
Plan to Share IPD: No